CLINICAL TRIAL: NCT03252782
Title: Three Dimensional Stereophotogrammetric Comparison of Intraoral Maxillary Molar Distalization and Functional Mandibular Advancement on Facial Soft Tissues
Brief Title: Comparison of Distalization and Functional Appliance Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Asli Baysal, Associate Professor, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-TDU-DİŞF-0023
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Mandibular Retrognathism
Keywords: Soft Tissue; Functional Appliance; Maxillary Molar Distalization
MeSH Terms: interventions — Orthodontic Appliances, Functional

STUDY DESIGN:
Intervention Model Description: 2-arm parallel-group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Treatment (Active Comparator): Acrylic Splint Herbst Appliance
  Interventions: Device: Herbst Appliance
- Distalization Treatment (Active Comparator): Mini-implant-borne Distal Jet Appliance
  Interventions: Device: Distal Jet Appliance

INTERVENTIONS:
Device: Herbst Appliance — Acrylic Splint Herbst Appliance
  Arms: Functional Treatment
Device: Distal Jet Appliance — Anterior Median Palate Implant Borne Distal Jet Appliance
  Arms: Distalization Treatment

SUMMARY:
The correction of Class II malocclusion is one of the most common problems facing the orthodontist, with an estimated one-third of all orthodontic patients treated for this condition. Many strategies are available for Class II treatment on growing patients, and most orthodontists tend to choose a treatment protocol based on what part of the craniofacial deformity they believe the appliance will affect the most. A number of authors have described the dentoalveolar and skeletal changes induced by the Herbst appliance. The dentoalveolar effects consist of distalization of the maxillary molars and forward movement of the mandibular dentition. The main skeletal change "mandibular stimulation" is acceleration of a patient's inherent mandibular growth rather than increased growth beyond what would occur without treatment. Maxillary molar distalization, is one of the Class II treatment. Mini-implants have become popular in recent years, and various kinds of mini-implant-borne distalization approaches have been described. Because Class II correction appears to be achievable with either appliance, a follow-up question is whether there is a difference in the esthetic outcomes. However, because of the complexity of the human face and the subjectivity of facial beauty, a simple set of measures of lines or angles cannot quantify facial beauty. With the advances in 3-dimensional imaging, it is now possible to capture and superimpose digital images and measure the changes in the soft tissues from 3-dimensional images. Such advances in facial imaging allow a more thorough investigation of changes in 3 dimensions and prevent the inherent loss of information that results from 2-dimensional imaging. Optical scanners with short shutter speeds are convenient for clinicians and patients for capturing soft-tissue records. Bearing in mind that the aim of orthodontic treatment is to achieve facial harmony along with excellent occlusion, one of the most important objectives of an orthodontist should be the improvement of facial appearance. Therefore, it is important to gain a better understanding of how or whether orthodontic procedures affect the appearance of the soft tissues. Thus, the aim of this clinical trial is three dimensional evaluation of soft tissue facial changes on late mixed dentition patients following maxillary arch distalization with palatal screws one group and acrylic split herbst patients on other group and to compare these changes.

DETAILED DESCRIPTION:
The correction of Class II malocclusion is one of the most common problems facing the orthodontist, with an estimated one-third of all orthodontic patients treated for this condition.

Many strategies are available for Class II treatment on growing patients, and most orthodontists tend to choose a treatment protocol based on what part of the craniofacial deformity they believe the appliance will affect the most.

A number of authors have described the dentoalveolar and skeletal changes induced by the Herbst appliance. The dentoalveolar effects consist of distalization of the maxillary molars and forward movement of the mandibular dentition. The main skeletal change "mandibular stimulation" is acceleration of a patient's inherent mandibular growth rather than increased growth beyond what would occur without treatment.

Maxillary molar distalization, is one of the Class II treatment. Mini-implants have become popular in recent years, and various kinds of mini-implant-borne distalization approaches have been described.

Because Class II correction appears to be achievable with either appliance, a follow-up question is whether there is a difference in the esthetic outcomes. However, because of the complexity of the human face and the subjectivity of facial beauty, a simple set of measures of lines or angles cannot quantify facial beauty.

Being the principle quantifiable diagnostic tool, the use of lateral head films lead orthodontists to have thought primarily in two dimensions. With the advances in 3-dimensional imaging, it is now possible to capture and superimpose digital images and measure the changes in the soft tissues from 3-dimensional images. Such advances in facial imaging allow a more thorough investigation of changes in 3 dimensions and prevent the inherent loss of information that results from 2-dimensional imaging. Optical scanners with short shutter speeds are convenient for clinicians and patients for capturing soft-tissue records.

Bearing in mind that the aim of orthodontic treatment is to achieve facial harmony along with excellent occlusion, one of the most important objectives of an orthodontist should be the improvement of facial appearance. Therefore, it is important to gain a better understanding of how or whether orthodontic procedures affect the appearance of the soft tissues. Thus, the aim of this clinical trial is three dimensional evaluation of soft tissue facial changes on late mixed dentition patients following maxillary arch distalization with palatal screws one group and acrylic split herbst patients on other group and to compare these changes.

ELIGIBILITY:
Inclusion Criteria:

Angle Class II molar relation, Skeletal Class II depends on mandibular retrognathia , Crowding less than 4 mm, Normal growth pattern, No systematic or oral disease, No previous orthodontic treatment

Exclusion Criteria:

Missing teeth, Severe facial asymmetry, Poor oral hygiene

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Soft Tissue Difference | Estimated 1 year
  Three-Dimensional Soft Tissue Changes Before and After Treatment